CLINICAL TRIAL: NCT03564158
Title: A Randomized, Placebo- and Positive-Controlled, Crossover Study to Evaluate the Effect of Meropenem-Vaborbactam on the QT/QTc Interval in Healthy Volunteers
Brief Title: Evaluate Effects of Meropenem-Vaborbactam on QT/QTc in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rempex (a wholly owned subsidiary of Melinta Therapeutics, Inc.) (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: Rempex 512
Record Dates: First submitted 2018-04-30; First posted 2018-06-20 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Healthy
MeSH Terms: interventions — meropenem and vaborbactam; Sodium Chloride; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only Moxifloxacin will be administered open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- meropenem 2 g- vaborbactam 2 g (Experimental): Approved Dose
  Interventions: Drug: meropenem-vaborbactam
- meropenem-vaborbactam (dose TBD) (Experimental): Supratherapeutic Dose
  Interventions: Drug: meropenem-vaborbactam
- Moxifloxacin 400 mg (Active Comparator): Active Control
  Interventions: Drug: Moxifloxacin
- Normal Saline (placebo) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: meropenem-vaborbactam — Meropenem-Vaborbactam being studied for effects on TQT
  Other Names: Vabomere
  Arms: meropenem 2 g- vaborbactam 2 g; meropenem-vaborbactam (dose TBD)
Drug: Placebo — Placebo
  Other Names: Saline
  Arms: Normal Saline (placebo)
Drug: Moxifloxacin — Active Comparator
  Other Names: Moxi
  Arms: Moxifloxacin 400 mg

SUMMARY:
This Thorough-QT (TQT) study in healthy volunteers will be conducted in two phases. Phase One will be used to identify a safe supratherapeutic dose to be used in the TQT study (Phase Two). Phase Two will be a 4-way crossover TQT study. Thirty-two subjects will receive all 4 of the following treatments in randomized sequence.

1. meropenem-vaborbactam 4 g (meropenem 2 g- vaborbactam 2 g) therapeutic dose infused intravenously over 3 hours
2. meropenem-vaborbactam supratherapeutic dose to be determined infused intravenously over 3 hours.
3. Placebo (normal saline) to match meropenem-vaborbactam volume infusion over 3 hours
4. Moxifloxacin 400 mg positive control (oral; open-label)

DETAILED DESCRIPTION:
This Thorough-QT (TQT) study in healthy volunteers will be conducted in two phases. Phase One (n=15) will be used to identify a safe supratherapeutic dose to be used in the TQT study (Phase Two). Phase Two will be a randomized, placebo and positive-controlled, 4-way crossover TQT study. Thirty-two subjects will receive all 4 of the following treatments in randomized sequence.

1. meropenem-vaborbactam 4 g (meropenem 2 g- vaborbactam 2 g) therapeutic dose infused intravenously over 3 hours
2. meropenem-vaborbactam supratherapeutic dose to be determined infused intravenously over 3 hours.
3. Placebo (normal saline) to match meropenem-vaborbactam volume infusion over 3 hours
4. Moxifloxacin 400 mg positive control (oral; open-label)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject between 18 and 55 years of age, inclusive, with a body mass index (BMI) ≥18 to ≤33 kilogram (kg)/m2.
2. All women of child-bearing potential must agree to use an adequate method of contraception during the study and for 30 days after the last dose. Accepted methods of contraception include: mechanical products (e.g., intrauterine device) or double-barrier methods (e.g., diaphragm, condoms, cervical cap) with spermicide or hormonal contraceptives (i.e., oral, implanted or injectable contraceptive hormones) or abstinence. Oral contraceptives must be used together with a second method of birth control. If the female subject has a male partner who has had a vasectomy, one additional form of medically acceptable contraception (condom or spermicide) must also be used. The subject's understanding of this requirement must be documented by the Investigator.

   Males with female partners of childbearing potential must agree to use a highly effective, medically acceptable form of contraception from the Screening period through 30 days after the last dose. Males with female partners of childbearing potential who themselves are surgically sterile (status post vasectomy) must agree to use condoms with spermicide over the same period of time. Male subjects must agree to practice the above birth control methods for 30 days after the final dose. Males must agree to not donate sperm through 30 days after the final dose.
3. Stable health based on no clinically-significant findings on the medical history, physical examination, or clinical laboratory test results at screening and prior to study drug administration (as determined and documented by the Investigator).
4. Willing to comply with all study activities and procedures and provides written informed consent prior to any study procedures

Exclusion Criteria:

1. Known hypersensitivity to beta-lactam antibiotics (including meropenem), fluoroquinolone antibiotics (including moxifloxacin) or vaborbactam.
2. An uninterpretable or abnormal screening electrocardiogram (ECG) indicating a second or third degree atrioventricular block, or any rhythm other than sinus rhythm that is interpreted by the investigator to be clinically significant or one or more of the following: QRS interval >110 milliseconds (ms); QTcF >430 ms (males) and >450 ms (females); PR interval >200 ms; heart rate (HR) <50 beats per minutes (bpm); or >90 bpm.
3. History of risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina. Subjects will also be excluded if there is a family history of long QT syndrome or Brugada syndrome or unexplained sudden death.
4. Subject has any clinically relevant abnormalities, as determined by the Investigator, in the laboratory results at Screening or admission of each study period
5. Serum potassium, serum magnesium, or albumin-corrected calcium lower than the lower limit of normal for the reference lab at Screening or admission of each study period. Calcium will be corrected for albumin using the formula: Corrected Calcium = (0.8 * (Normal Albumin - Pt's Albumin)) + Serum Ca where Normal Albumin is 4.0 g/dL.
6. Hemoglobin and hematocrit lower than the lower limit of normal for the reference lab at Screening.
7. Subject has an abnormal liver function tests: alanine aminotransferase [ALT], aspartate aminotransferase [AST], or bilirubin greater than 1.2X the upper limits of normal at Screening.
8. History of central nervous system (CNS) disorder including convulsions.
9. A sustained supine systolic blood pressure >140 mmHg or <90 mmHg or a supine diastolic blood pressure >90 mmHg or <50 mmHg at Screening or Check in (Day -1). Blood pressure may be retested once in the supine position. The blood pressure abnormality is considered sustained if either the systolic or the diastolic pressure values are outside the stated limits after 2 assessments, in which case the subject should not be randomized.
10. Impaired renal function as evidenced by estimated glomerular filtration rate (eGFR) <50.
11. Unstable cardiovascular disease, including recent myocardial infarction or cardiac arrhythmia.
12. History of acquired immunodeficiency syndrome or history of a positive test result for human immunodeficiency virus (HIV), hepatitis C virus (HCV) antibody, or hepatitis B surface antigen (HBsAg) at Screening.
13. Positive drug, alcohol, or tobacco screen.
14. Clinically-significant illness, including viral syndromes within 3 weeks of dosing.
15. Women who are pregnant (or planning to become pregnant within the next 6 months) or currently breastfeeding. A negative serum pregnancy test is required before enrolling in the study.
16. Participation in another investigational drug or device study or treated with an investigational drug within 30 days or 5 half lives, whichever is longer, before dosing. Any subject who participated in Phase One of this trial is not eligible to participate in Phase Two.
17. Consumed more than 28 units of ethanol per week at any time in the 6 months before dosing (1 unit of ethanol is equivalent to 8 ounces of beer, 4 ounces of wine, or 1 ounce of spirits) or history of alcoholism and/or drug/chemical abuse.
18. Use of prescription medications (with the exception of oral contraceptives and hormone replacement therapy), including nonsteroidal anti-inflammatory drugs or sucralfate and medications known to prolong the QT/QTc interval or natural health products/herbal preparations within 14 days or 5 half lives (whichever is longer) before study drug dosing, or use of an over-the-counter (OTC) medication (excluding acetaminophen), vitamins, or supplements (including omega-3 fish oils) within 7 days before study drug dosing.
19. Use of alcohol , caffeine , or xanthine containing products, Seville oranges (sour), grapefruit, or grapefruit juice, within 72 hours before study drug dosing.
20. Current use or has used tobacco- or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.) 30 days before study drug dosing.
21. Strenuous activity (e.g., sports) from 96 hours (4 days) prior to entry into the clinical research unit and throughout the study (until the final follow-up call is conducted).
22. Donated more than 500 milliliter (mL) of blood or significant blood loss within 60 days prior to signing the informed consent form.
23. Any other medical, psychological, or social condition that, in the opinion of the principal investigator or the medical monitor, would prevent the subject from fully participating in the study, would represent a concern for study compliance, or would constitute a safety concern to the subject.
24. An employee of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as a family member of the employee or investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change-from-baseline QTcF interval (ΔΔQTcF) | 24 hours after start of dosing
  Change in placebo corrected QTcF after dosing

SECONDARY OUTCOMES:
Change-from-baseline HR | 24 hours after start of dosing
  Change in HR after dosing
Change-from-baseline QTcF inteval | 24 hours after start of dosing
  Change in QTcF after dosing
Change-from-baseline PR interval | 24 hours after start of dosing
  Change in PR after dosing
Change-from-baseline QRS interval | 24 hours after start of dosing
  Change in QRS after dosing
Change-from-baseline RR interval | 24 hours after start of dosing
  Change in RR after dosing
Change-from-baseline QT interval | 24 hours after start of dosing
  Change in QT interval after dosing

OTHER OUTCOMES:
Number of participants with treatment emergent adverse events as assessed by CTCAE v4.3 | 7 days after treatment
  Safety evaluation (non-serious Treatment Emergent Adverse Events) of high dose of meropenem-vaborbactam
Number of participants with treatment emergent serious adverse events as assessed by CTCAE v4.3. | 7 days after treatment
  Safety evaluation (serious Treatment Emergent Adverse Event) of high dose of meropenem-vaborbactam

CONTACTS AND LOCATIONS:
Overall Officials: Sue Cammarata, Study Director — Melinta Therapeutics, Inc.
Locations (1):
- Pharmaron Cpc, Inc, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No